CLINICAL TRIAL: NCT00282542
Title: The Use of Human Hepatocyte Transplantation as a Life Support Bridge in Terminal Liver Failure
Brief Title: Hepatocyte Transplantation as a Life Support Bridge
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCU124
Record Dates: First submitted 2006-01-20; First posted 2006-01-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Fulminant Liver Failure
Keywords: Hepatocytes
MeSH Terms: conditions — Liver Failure, Acute

INTERVENTIONS:
Procedure: Hepatocyte Infusion

SUMMARY:
The purpose of this study is to gain knowledge about the result of infusing liver cells, carefully matched to blood type, into a subject's body. The hope is that this procedure will aid functions of the liver and prevent death, enable a transplant procedure to be carried out if a donated liver becomes available, and lessen complications in postoperative recovery. There is no guarantee that any of these benefits will be re eived, but even if they are not, the hope is that knowledge gained by using this procedure will be of future benefit to others who also suffer from liver disease.

DETAILED DESCRIPTION:
Adult and pediatric patients eligible for liver transplantation who require intensive care unit admission for multisystem organ failure in addition to liver failure, without systemic sepsis, are eligible for liver cell transplantation regardless of race, sex or financial support.

Failure of 3 or more organ systems are the criterion used to select patients with as close to 100% mortality as possible without solid organ transplant.

Hepatocytes, isolated from excess liver tissure from reduced liver transplant procedures or from donor livers not used for transplantation, are prepared by a complex process and then are infused, guided by radiology into the splenic artery or portal vein of the patient. Patients must be on immunosuppression therapy for as long as the hepatocytes are living and beneficial to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to VCU Health System ICU in fulminant Liver Failure in addition to multisystem organ failure

Exclusion Criteria: Patients with Sepsis

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-05; Study Completion 2006-01

PRIMARY OUTCOMES:
Survival to liver transplantation

SECONDARY OUTCOMES:
Liver Function Normalization

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Fisher, MD, FACS, Principal Investigator — VCU Health System